CLINICAL TRIAL: NCT04194814
Title: Validation of a Novel Composite of Skin Biomarkers as a Primary Outcome Measure for Evaluating the Safety of Treatments for Atopic Dermatitis: a Randomized Controlled Trial (Phase 2) Comparing the Effects of Crisaborole 2% Ointment to Betamethasone Valerate 0.1% Cream on Skin Structure and Function in Participants With Atopic Dermatitis.
Brief Title: Skin bioMARkers for Atopic Eczema Therapy Evaluation
Acronym: SMART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STH19966; 2019-002643-23 (EudraCT Number); WI242083-UK [Eucrisa] (Other Grant/Funding Number: Pfizer, Inc.); 269415 (Other: IRAS)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Atopic Eczema/Dermatitis (Non-Specific)
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — crisaborole; Ointments; Betamethasone Valerate

STUDY DESIGN:
Intervention Model Description: An observer-blind forearm-controlled clinical trial in 37 AD patients, wherein each participant will undergo 4 weeks treatment with crisaborole (2%) ointment on one forearm and betamethasone valerate (0.1%) cream on the other (twice daily application in each case and randomised site allocation). At the start of the study the skin of the test sites (forearms) will be clear of the signs of AD so that the investigation focuses on local adverse effects on the skin as opposed to anti-inflammatory effects (focus on local adverse effects and not clinical efficacy). The condition of the skin will be assessed before, during and after treatment.
Masking Description: Allocation of the treatments to the test sites (right/left forearm) will be randomised (to avoid site position-dependent artefacts) Observer-blind - The collection of study data will be conducted in a separate area (dedicated skin barrier research suite) by a separate team (comprising skilled dermatology researchers) who will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- crisaborole and topical Corticosteroid (Other): crisaborole (2%) ointment on the other forearm, twice daily application for 4 weeks (randomised site allocation)
  betamethasone valerate (0.1%) cream on one forearm, twice daily application for 4 weeks (randomised site allocation)
  Interventions: Drug: crisaborole (2%) ointment; Drug: betamethasone valerate 0.1% cream

INTERVENTIONS:
Drug: crisaborole (2%) ointment — twice daily application on one forearm for 4 weeks (randomised site allocation)
  Other Names: Eucrisa
Drug: betamethasone valerate 0.1% cream — twice daily application on one forearm for 4 weeks (randomised site allocation)
  Other Names: Betnovate cream

SUMMARY:
The study aims to investigate two new non-invasive technologies for assessing skin properties to identify and validate a range of safety biomarkers that may be considered useful as primary outcome measures for evaluating the safety of topical treatments in atopic dermatitis. The method of assessing these biomarker technologies will be to determine whether twice daily treatment with crisaborole (2%) ointment, compared to betamethasone valerate (0.1%) cream, for up to 4 weeks, may cause skin structure or function changes, like skin atrophy, in patients with atopic dermatitis (AD).

DETAILED DESCRIPTION:
The first-line drug treatment for mild-moderate AD are currently topical corticosteroids (TCS) with recognized efficacy. However, their prolonged or inappropriate use, can lead to local adverse effects. Side-effects of topical corticosteroids comprise a variety of skin changes in the sense of skin atrophy thinning of the skin and in some cases development of telangiectasia, spontaneous scars, folliculitis, striae distensae (stretch marks), contact dermatitis, acne or rosacea depending on potency, galenic formulation, patient age and body area to which the medication will be applied, exposure time.

Assessing the safety (local adverse effects) of current or new treatments and new treatment approaches using existing treatments through noninvasively monitor on possible early skin (subclinical) changes associated with the local clinical adverse effects of treatment may be an effective step for an enhanced AD treatment management.

Primary Aim: To further develop and validate two new non-invasive technologies for the assessment of early sub-clinical skin changes associated with adverse effects and to derive an optimum panel of safety biomarkers for use in future clinical trials of topical anti-inflammatory treatments.

The safety of two topical anti-inflammatory treatments for AD will be compared in this clinical trial, with a focus on early sub-clinical signs: crisaborole 2% ointment and betamethasone valerate 0,1% cream. Step 1 involves the collection of data on the early sub-clinical skin changes using the non-invasive technologies: OCT and FTIR spectroscopy. The data from this study will then be used to identify and refine biophysical biomarkers of skin atrophy and skin barrier disruption in steps 2 and 3.

Secondary Aim: To determine the relative local skin effects of crisaborole (2%) ointment compared to a potent and moderately potent TCS in participants with mild to moderate AD. The focus is on 'early biomarkers' of 'local skin changes'and not clinical efficacy, which has been established in previous trials.

Rationale for selecting the two comparators are related to prescription behaviors in UK (Betamethasone valerate 0,1% cream) and with no reported TCS-like local adverse effects profile (crisaborole 2% ointment)

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with AD defined according to the UK working party diagnostic criteria
* Male or female aged 18-65 years old at baseline (Visit 1)
* Volunteer understands the purpose, modalities and potential risk of the trial
* Participants able to read and understand English
* Participants willing to sign the informed consent

Exclusion Criteria:

* Participants with a known allergy/hypersensitivity to any of the excipients of the trial preparations.
* Participants with acne, suntan, birth marks, multiple nevi, tattoos, blemishes or dense body hair that obstruct the test areas.
* Investigator assessment of eczema severity at the treatment (anatomical) sites is almost clear or greater (score ≥1) based on the Investigators static global assessment scale at screening and baseline. At the start of the study the skin of the test sites (forearms) will therefore be clear (0) of the signs of eczema
* Participants with a condition that in the opinion of the investigator contradicts participation in the study.
* Pregnant female participants; breastfeeding female participants; and female participants of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Use of any topical product on the test areas within 7 days prior to Baseline/Day 1, including cosmetic moisturizers and sunscreen. Participants using any topical products on the test areas within 7 days at the screening visit will be eligible if they are willing and able to wash-out these products for 7 days in total and for the duration of the trial. Such participants will be potentially eligible at screening and will be confirmed as eligible if adequate washout is confirmed at visit 1. Use of moisturizers and/or sunscreen is permitted during the study to manage dry skin and sun exposure in areas surrounding but not on or overlapping the test areas.
* Participants who have used a tanning bed within 28 days of baseline (visit 1). Participants who have used a sunbed within 28 days at the screening visit will be eligible if they are willing and able to wash-out for 28 days in total and for the duration of the trial. Such participants will be potentially eligible at screening and will be confirmed as eligible if adequate washout is confirmed at visit 1.
* Participants who have used any medication that could interfere with the trial aim prior to the start of the study (baseline/visit 1). Participants using such medication at the screening visit will be eligible if they are willing and able to wash-out these treatments for the applicable washout period as defined by in section 8.8 'Prior and Concomitant Medication' and for the duration of the trial. Such participants will be potentially eligible at screening and will be confirmed as eligible if adequate washout is confirmed at visit 1.
* Participants currently participating in another interventional clinical trial.
* Volunteer is incapable of giving fully informed consent.
* Participants judged by the PI to be inappropriate for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cork, MB.ChB, Principal Investigator — The University of Sheffield & Sheffield Teaching Hospitals NHS FT
Locations (1):
- Sheffield Dermatology Research, University of Sheffield Medical School, The Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Odhiambo JA, Williams HC, Clayton TO, Robertson CF, Asher MI; ISAAC Phase Three Study Group. Global variations in prevalence of eczema symptoms in children from ISAAC Phase Three. J Allergy Clin Immunol. 2009 Dec;124(6):1251-8.e23. doi: 10.1016/j.jaci.2009.10.009. PMID 20004783
- [Background] Kerr OA, Tidman MJ, Walker JJ, Aldridge RD, Benton EC. The profile of dermatological problems in primary care. Clin Exp Dermatol. 2010 Jun;35(4):380-3. doi: 10.1111/j.1365-2230.2009.03586.x. Epub 2009 Oct 23. PMID 19874334
- [Background] Cork MJ, Danby SG, Vasilopoulos Y, Hadgraft J, Lane ME, Moustafa M, Guy RH, Macgowan AL, Tazi-Ahnini R, Ward SJ. Epidermal barrier dysfunction in atopic dermatitis. J Invest Dermatol. 2009 Aug;129(8):1892-908. doi: 10.1038/jid.2009.133. Epub 2009 Jun 4. PMID 19494826
- [Background] Punekar YS, Sheikh A. Establishing the sequential progression of multiple allergic diagnoses in a UK birth cohort using the General Practice Research Database. Clin Exp Allergy. 2009 Dec;39(12):1889-95. doi: 10.1111/j.1365-2222.2009.03366.x. Epub 2009 Oct 7. PMID 19817751
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Lewis-Jones S, Mugglestone MA; Guideline Development Group. Management of atopic eczema in children aged up to 12 years: summary of NICE guidance. BMJ. 2007 Dec 15;335(7632):1263-4. doi: 10.1136/bmj.39405.503773.AD. No abstract available. PMID 18079551
- [Background] Hengge UR, Ruzicka T, Schwartz RA, Cork MJ. Adverse effects of topical glucocorticosteroids. J Am Acad Dermatol. 2006 Jan;54(1):1-15; quiz 16-8. doi: 10.1016/j.jaad.2005.01.010. PMID 16384751
- [Background] Schmitt J, von Kobyletzki L, Svensson A, Apfelbacher C. Efficacy and tolerability of proactive treatment with topical corticosteroids and calcineurin inhibitors for atopic eczema: systematic review and meta-analysis of randomized controlled trials. Br J Dermatol. 2011 Feb;164(2):415-28. doi: 10.1111/j.1365-2133.2010.10030.x. Epub 2010 Nov 23. PMID 20819086
- [Background] Batchelor JM, Ridd MJ, Clarke T, Ahmed A, Cox M, Crowe S, Howard M, Lawton S, McPhee M, Rani A, Ravenscroft JC, Roberts A, Thomas KS. The Eczema Priority Setting Partnership: a collaboration between patients, carers, clinicians and researchers to identify and prioritize important research questions for the treatment of eczema. Br J Dermatol. 2013 Mar;168(3):577-82. doi: 10.1111/bjd.12040. Epub 2013 Jan 18. PMID 22963149
- [Background] Byers RA, Maiti R, Danby SG, Pang EJ, Mitchell B, Carre MJ, Lewis R, Cork MJ, Matcher SJ. Sub-clinical assessment of atopic dermatitis severity using angiographic optical coherence tomography. Biomed Opt Express. 2018 Mar 29;9(4):2001-2017. doi: 10.1364/BOE.9.002001. eCollection 2018 Apr 1. PMID 29675335
- [Background] Ugryumova N, Jacobs J, Bonesi M, Matcher SJ. Novel optical imaging technique to determine the 3-D orientation of collagen fibers in cartilage: variable-incidence angle polarization-sensitive optical coherence tomography. Osteoarthritis Cartilage. 2009 Jan;17(1):33-42. doi: 10.1016/j.joca.2008.05.005. Epub 2008 Jul 14. PMID 18621555
- [Background] Danby SG, Brown K, Higgs-Bayliss T, Chittock J, Albenali L, Cork MJ. The Effect of an Emollient Containing Urea, Ceramide NP, and Lactate on Skin Barrier Structure and Function in Older People with Dry Skin. Skin Pharmacol Physiol. 2016;29(3):135-47. doi: 10.1159/000445955. Epub 2016 Jun 2. PMID 27251427
- [Background] Boncheva M, Damien F, Normand V. Molecular organization of the lipid matrix in intact Stratum corneum using ATR-FTIR spectroscopy. Biochim Biophys Acta. 2008 May;1778(5):1344-55. doi: 10.1016/j.bbamem.2008.01.022. Epub 2008 Feb 11. PMID 18298945
- [Background] Damien F, Boncheva M. The extent of orthorhombic lipid phases in the stratum corneum determines the barrier efficiency of human skin in vivo. J Invest Dermatol. 2010 Feb;130(2):611-4. doi: 10.1038/jid.2009.272. Epub 2009 Sep 3. No abstract available. PMID 19727117
- [Background] Chittock J, Brown K, Cork MJ, Danby SG. Comparing the Effect of a Twice-weekly Tacrolimus and Betamethasone Valerate Dose on the Subclinical Epidermal Barrier Defect in Atopic Dermatitis. Acta Derm Venereol. 2015 Jul;95(6):653-8. doi: 10.2340/00015555-2048. PMID 25594610
- [Background] Danby SG, Chittock J, Brown K, Albenali LH, Cork MJ. The effect of tacrolimus compared with betamethasone valerate on the skin barrier in volunteers with quiescent atopic dermatitis. Br J Dermatol. 2014 Apr;170(4):914-21. doi: 10.1111/bjd.12778. PMID 24328907
- [Background] Kezic S, O'Regan GM, Yau N, Sandilands A, Chen H, Campbell LE, Kroboth K, Watson R, Rowland M, McLean WH, Irvine AD. Levels of filaggrin degradation products are influenced by both filaggrin genotype and atopic dermatitis severity. Allergy. 2011 Jul;66(7):934-40. doi: 10.1111/j.1398-9995.2010.02540.x. Epub 2011 Jan 25. PMID 21261659
- [Background] Lu Z, Kasaragod D, Matcher SJ. Conical scan polarization-sensitive optical coherence tomography. Biomed Opt Express. 2014 Feb 18;5(3):752-62. doi: 10.1364/BOE.5.000752. eCollection 2014 Mar 1. PMID 24688811
- [Background] Chittock J, Cooke A, Lavender T, Brown K, Wigley A, Victor S, Cork MJ, Danby SG. Development of stratum corneum chymotrypsin-like protease activity and natural moisturizing factors from birth to 4 weeks of age compared with adults. Br J Dermatol. 2016 Oct;175(4):713-20. doi: 10.1111/bjd.14568. Epub 2016 Jul 22. PMID 26994359
- [Background] Danby SG, AlEnezi T, Sultan A, Lavender T, Chittock J, Brown K, Cork MJ. Effect of olive and sunflower seed oil on the adult skin barrier: implications for neonatal skin care. Pediatr Dermatol. 2013 Jan-Feb;30(1):42-50. doi: 10.1111/j.1525-1470.2012.01865.x. Epub 2012 Sep 20. PMID 22995032
- [Background] Brancaleon L, Bamberg MP, Sakamaki T, Kollias N. Attenuated total reflection-Fourier transform infrared spectroscopy as a possible method to investigate biophysical parameters of stratum corneum in vivo. J Invest Dermatol. 2001 Mar;116(3):380-6. doi: 10.1046/j.1523-1747.2001.01262.x. PMID 11231311
- [Background] Ring A, Schreiner V, Wenck H, Wittern KP, Kupper L, Keyhani R. Mid-infrared spectroscopy on skin using a silver halide fibre probe in vivo. Skin Res Technol. 2006 Feb;12(1):18-23. doi: 10.1111/j.0909-725X.2006.00130.x. PMID 16420534
- [Background] Cooke A, Cork MJ, Victor S, Campbell M, Danby S, Chittock J, Lavender T. Olive Oil, Sunflower Oil or no Oil for Baby Dry Skin or Massage: A Pilot, Assessor-blinded, Randomized Controlled Trial (the Oil in Baby SkincaRE [OBSeRvE] Study). Acta Derm Venereol. 2016 Mar;96(3):323-30. doi: 10.2340/00015555-2279. PMID 26551528
- [Background] Kao JS, Fluhr JW, Man MQ, Fowler AJ, Hachem JP, Crumrine D, Ahn SK, Brown BE, Elias PM, Feingold KR. Short-term glucocorticoid treatment compromises both permeability barrier homeostasis and stratum corneum integrity: inhibition of epidermal lipid synthesis accounts for functional abnormalities. J Invest Dermatol. 2003 Mar;120(3):456-64. doi: 10.1046/j.1523-1747.2003.12053.x. PMID 12603860
- See also: Atopic eczema in children - Guideline consultation: National Institute for Clinical Excellence, Department of Health, UK — https://www.nice.org.uk/guidance/cg57/resources/atopic-eczema-in-under-12s-diagnosis-and-management-pdf-975512529349
- See also: Danby SG, Wan H, Chittock J et al. Characterisation of the skin barrier defect in atopic dermatitis using in vivo ATR-FTIR molecular spectroscopy. J Invest Dermatol 2016; 136: S182. — https://static1.squarespace.com/static/5f660d2b22e95f46e1f67c92/t/5f873e1cfaba973d5cdf13c1/1602698786483/B.pdf
- See also: Lu Z, et al. Optical coherence tomography demonstrates differential epidermal thinning of human forearm volar skin after 2 weeks application of a topical corticosteroid vs a non-steroidal anti-inflammatory alternative. Proc. SPIE 2013; 85 — https://www.spiedigitallibrary.org/conference-proceedings-of-spie/8565/1/Optical-coherence-tomography-demonstrates-differential-epidermalthinning-of-human-forearm-volar/10.1117/12.2006104.full
- See also: Takada S, Naito S, Sonoda J et al. Noninvasive In Vivo Measurement of Natural Moisturizing Factor Content in Stratum Corneum of Human Skin by Attenuated Total Reflection Infrared Spectroscopy. Applied Spectroscopy 2012; 66: 26-32. — https://www.osapublishing.org/as/abstract.cfm?uri=as-66-1-26

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 20/11/2020 and ended 27/07/2021. 37 participants were recruited.
  Recruitment was conducted by the Sheffield Dermatology Research Group in several ways:
  General advertisement using posters. Email lists. Outpatient contact including local GP practices.
Pre-assignment Details: Some participants, who were currently using treatments for eczema, needed to undergo a 'wash out' period, where the use of these treatments was stopped, prior to the first study visit. The duration of the wash-out depended on the type of treatment, and varied from 7 days for emollients to 12 weeks for intravenous biologic therapies.
Groups:
- Betamethasone Valerate (0.1%) Cream LEFT/Crisaborole (2%) Ointment RIGHT: All participants who treated the left forearm with Betamethasone valerate (0.1%) cream and the right forearm with Crisaborole (2%) ointment. Twice daily application for 4 weeks (randomised site allocation).
- Crisaborole (2%) Ointment LEFT/Betamethasone Valerate (0.1%) Cream RIGHT: All participants who treated the left forearm with Crisaborole (2%) ointment and the right forearm with Betamethasone valerate (0.1%) cream. Twice daily for 4 weeks (randomised site allocation).
Period: Overall Study
Arm/Group | Betamethasone Valerate (0.1%) Cream LEFT/Crisaborole (2%) Ointment RIGHT | Crisaborole (2%) Ointment LEFT/Betamethasone Valerate (0.1%) Cream RIGHT
Started | 18 | 19
Completed | 15 | 17
Not Completed | 3 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled: All enrolled participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 37
Atopic dermatitis as defined by UK working party diagnostic criteria [Count of Participants; unit: Participants] | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Epidermal Thickness
Description: The difference in the change in epidermal thickness, measured by structural OCT, between the sites treated with crisaborole (2%) ointment and betamethasone valerate (0.1%) cream.
Time Frame: Day 1 - Day 57
Measure: Mean (95% Confidence Interval); unit: µm
Groups:
- Betamethasone Valerate (0.1%) Cream: All sites (left or right) treated with Betamethasone valerate (0.1%) cream.
- Crisaborole (2%) Ointment: All sites (left or right) treated with Crisaborole (2%) ointment.
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
µm
  Day 1 to Day 29 | -31.66 [-35.31 to -28.01] | -13.76 [-17.42 to -10.10]
  Day 1 to Day 15 | -28.65 [-31.58 to -25.73] | -14.41 [-17.35 to -11.48]
  Day 29 to Day 57 | 24.94 [21.39 to 28.5] | 11.63 [8.07 to 15.19]

2. Secondary Outcome: Analysis of Change in Objective Erythema
Description: Analysis of the difference in the change in skin redness/erythema (relating to tolerability) during and after 28 days treatment determined by Mexameter measured on day 1, day 15, day 29 and day 57.
  The Mexameter device has a range of 0-999AU (arbitrary units) and the lower the value, the better the condition of the skin. Objective redness can be classified using the following scale: 0-170AU - No erythema; 170-330AU - Minimal erythema; 330-450AU - Diffuse erythema; 450-570AU - High erythema; over 570AU - Extreme erythema
Time Frame: Day 1, Day 15, Day 29 and Day 57
Population: 35 participants had complete data at Day 1. Each participant was expected to complete 56 days of treatment. A total of 5 participants were withdrawn before this point and so only 32 participants had data available for analysis at Day 29 and 57.
Measure: Mean (95% Confidence Interval); unit: AU
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
AU
  Baseline to Day 29: number analyzed (Participants) | 32 | 32
  Baseline to Day 29 | -27.61 [-43.48 to -11.73] | -1.16 [-17.04 to 14.72]
  Baseline to Day 15 | -45.04 [-59.08 to -31.01] | -23.61 [-37.65 to -9.57]
  Day 29 to Day 57 | 37.66 [22.80 to 52.51] | 2.84 [-12.02 to 17.69]

3. Secondary Outcome: TEWL - Skin Barrier Function
Description: Analysis of the change in Trans-Epidermal Water Loss (TEWL, relates to skin barrier function) during and after treatment. TEWL measurements on day 1, day 15, day 29 and day 57.
Time Frame: Day 1, Day 15, Day 29 and Day 57
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: g/m²/h
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
g/m²/h
  Baseline to Day 29: number analyzed (Participants) | 32 | 32
  Baseline to Day 29 | -0.52 [-1.62 to 0.59] | 2.06 [0.96 to 3.16]
  Baseline to Day 15 | -0.92 [-1.74 to -0.11] | 1.66 [0.85 to 2.48]
  Day 29 to Day 57: number analyzed (Participants) | 32 | 32
  Day 29 to Day 57 | 2.25 [0.79 to 3.72] | 0.21 [-1.26 to 1.67]

4. Secondary Outcome: TEWL - After Tape-stripping
Description: The difference in skin barrier integrity (TEWLts20) after 28 days treatment. TEWL measurements after tape-stripping (TEWLts20) on day 29
Time Frame: on Day 29, after 28 days treatment
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: g/m²/h
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
g/m²/h | 45.4 (23.01) | 34.1 (14.67)

5. Secondary Outcome: Comparison of TEWL - After Tape-stripping
Description: as for outcome 4
Time Frame: on Day 29, after 28 days treatment
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: g/m²/h
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
g/m²/h | 45.44 [37.14 to 53.74] | 34.13 [28.84 to 39.42]

6. Secondary Outcome: Skin Dryness
Description: The difference in the change in visual skin dryness during and after treatment. Visual skin dryness scored on day 1, day 15, day 29 and day 57. Visual skin dryness was scored using the following: 0 - Absent; 1 - Faint scaling, faint roughness and dull appearance; 2 - Small scales in combination with a few larger scales, slight roughness, whitish appearance; 3 - Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks; 4 - Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks. The lower the visual dryness score, the better the condition of the skin.
Time Frame: Visual skin dryness scored on day 1, day 15, day 29 and day 57
Population: Frequency of visual dryness scores on Day 1, Day 15, Day 29 and Day 57.
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 37 | 37
Participants
  Day 1: 0 | 36 | 35
  Day 1: 1 | 1 | 2
  Day 1: 2 | 0 | 0
  Day 15: number analyzed (Participants) | 35 | 35
  Day 15: 0 | 34 | 35
  Day 15: 1 | 1 | 0
  Day 15: 2 | 0 | 0
  Day 29: number analyzed (Participants) | 32 | 32
  Day 29: 0 | 30 | 31
  Day 29: 1 | 2 | 1
  Day 29: 2 | 0 | 0
  Day 57: number analyzed (Participants) | 32 | 32
  Day 57: 0 | 28 | 29
  Day 57: 1 | 3 | 2
  Day 57: 2 | 1 | 1

7. Secondary Outcome: Natural Moisturising Factor (NMF)
Description: The difference in Natural Moisturising Factor (NMF, filaggrin breakdown products) levels at the end of treatment.
  3 NMF components were measured: Urocanic acid (UCA), Pyrrolidone carboxylic acid (PCA) and Free amino acids (FAA) and are expressed together as total NMF (tNMF).
Time Frame: Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: moles/µg protein
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
moles/µg protein
  Total Natural Moisturising Factors (NMF) | 1.299 (0.6080) | 1.331 (0.5885)
  Pyrrolidone Carboxylic Acid (PCA) | 0.156 (0.844) | 0.157 (0.0708)
  Urocanic Acid (UCA) | 0.032 (0.0218) | 0.039 (0.0208)
  Free Amino Acids (FAA) | 1.111 (0.5164) | 1.135 (0.5215)

8. Secondary Outcome: Comparison of Natural Moisturising Factor (NMF) Between Treatments
Description: as for outcome 7
Time Frame: Day 29
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: nmoles/µg protein
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
nmoles/µg protein
  Total Natural Moisturising Factors (NMF) | 1.299 [1.080 to 1.518] | 1.331 [1.119 to 1.543]
  Pyrrolidone Carboxylic Acid (PCA) | 0.156 [0.125 to 0.186] | 0.157 [0.131 to 0.182]
  Urocanic Acid (UCA) | 0.032 [0.024 to 0.040] | 0.039 [0.031 to 0.046]
  Free Amino Acids (FAA) | 1.111 [0.925 to 1.297] | 1.135 [0.947 to 1.323]

9. Secondary Outcome: Change in Visual Redness/Erythema During and After 28 Days Treatment
Description: The difference in the change in visual skin redness during and after treatment. Visual skin redness scored on day 1, day 15, day 29 and day 57 by an experienced grader. Visual skin redness was scored using the following: 0 - No redness; 0.5/+ - Slight patchy erythema, barely perceptible; 1 - Slight uniform erythema, mild erythema; 2 - Moderate uniform erythema, moderate erythema; 3 - Strong erythema, marked erythema. The higher the visual redness score, the more inflamed the skin looks to the naked eye.
Time Frame: Visual skin redness scored on day 1, day 15, day 29 and day 57
Population: Frequency of visual dryness scores on Day 1, Day 15, Day 29 and Day 57.
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 37 | 37
Participants
  Day 1: 0 | 24 | 22
  Day 1: 0.5 | 13 | 15
  Day 1: 1 | 0 | 0
  Day 15: number analyzed (Participants) | 35 | 35
  Day 15: 0 | 26 | 24
  Day 15: 0.5 | 9 | 11
  Day 15: 1 | 0 | 0
  Day 29: number analyzed (Participants) | 32 | 32
  Day 29: 0 | 18 | 21
  Day 29: 0.5 | 11 | 9
  Day 29: 1 | 3 | 2
  Day 57: number analyzed (Participants) | 32 | 32
  Day 57: 0 | 16 | 20
  Day 57: 0.5 | 15 | 11
  Day 57: 1 | 1 | 1

10. Other Pre Specified Outcome: Superficial Plexus Depth
Description: The difference in the change in superficial plexus depth (μm) measured by angiographic OCT.
Time Frame: Day 1, Day 15, Day 29 and Day 57
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
µm
  Day 1 to Day 29: number analyzed (Participants) | 32 | 32
  Day 1 to Day 29 | -20.3 (17.44) | -9.5 (20.76)
  Day 1 to Day 15 | -22.3 (16.42) | -13.1 (19.11)
  Day 29 to Day 57: number analyzed (Participants) | 32 | 32
  Day 29 to Day 57 | 13.4 (20.60) | 7.3 (17.25)

11. Other Pre Specified Outcome: Blood Vessel Diameter
Description: The difference in the mean blood vessel diameter (μm) measured by angiographic OCT.
Time Frame: Day 1, Day 15, Day 29 and Day 57.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
µm
  Day 1 to Day 29: number analyzed (Participants) | 32 | 32
  Day 1 to Day 29 | -1.02 (4.432) | -1.04 (4.518)
  Day 1 to Day 15 | -0.37 (4.195) | -0.69 (3.964)
  Day 29 to Day 57: number analyzed (Participants) | 32 | 32
  Day 29 to Day 57 | 1.36 (3.320) | 0.13 (3.393)

12. Other Pre Specified Outcome: Blood Vessel Density
Description: The difference in the change in blood vessel density (segments/mm²) measured by angiographic OCT. Angiographic OCT images taken on Day 1, Day 15, Day 29 and Day 57.
Time Frame: Day 1, Day 15, Day 29 and Day 57.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: segments/mm²
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
segments/mm²
  Day 1 to Day 29: number analyzed (Participants) | 32 | 32
  Day 1 to Day 29 | -1.27 (18.381) | 3.37 (15.842)
  Day 1 to Day 15 | -1.12 (17.769) | -0.56 (16.825)
  Day 29 to Day 57: number analyzed (Participants) | 32 | 32
  Day 29 to Day 57 | 4.79 (17.677) | -0.15 (17.630)

13. Other Pre Specified Outcome: Collagen Matrix Index
Description: The difference in the change in collagen matrix index measured by polarisation sensitive (PS-)OCT. This metric relates to the arrangement and density of collagen fibres within the skin and is informed by birefringence data. Inhibition of collagen synthesis is an adverse effect associated with epidermal atrophy that occurs following long-term use of topical corticosteroids. There is no range for this measurement. The higher the level of change, the more damage has been done to the epidermis.
Time Frame: Day 1 and Day 29.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
AU | 100.0 (102.11) | -4.0 (78.55)

14. Other Pre Specified Outcome: Carboxylate 1 Levels
Description: The difference in the change in carboxylate 1 levels (indirect measure of NMF levels, not to be confused with direct quantification from stratum corneum samples by HPLC) in the stratum corneum measured by FTIR spectroscopy. FTIR spectra of the skin surface taken on Day 1, Day 15, Day 29 and Day 57.
  Carboxylate 1 is a component of Natural Moisturising Factors and relates to how well the skin retains water. There is no range for this measurement. The greater the value, the less able the skin is to hold onto water.
Time Frame: Day 1, Day 15, Day 29 and Day 57.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: absorbance units
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
absorbance units
  Day 1 to Day 29 | -6.75 (5.800) | -4.88 (5.450)
  Day 1 to Day 15 | -3.1 (4.887) | -3.52 (4.675)
  Day 29 to Day 57: number analyzed (Participants) | 31 | 31
  Day 29 to Day 57 | 6.97 (4.594) | 4.88 (4.686)

15. Other Pre Specified Outcome: Carboxylate 2 Levels
Description: The difference in the change in carboxylate 2 levels (indirect measure of NMF levels, not to be confused with direct quantification from stratum corneum samples by HPLC) in the stratum corneum measured by FTIR spectroscopy. FTIR spectra of the skin surface taken on Day 1, Day 15, Day 29 and Day 57.
  Carboxylate 2 is a component of Natural Moisturising Factors and relates to how well the skin retains water. There is no range for this measurement. The greater the value, the less able the skin is to hold onto water.
Time Frame: Day 1, Day 15, Day 29 and Day 57.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: absorbance units
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 35 | 35
absorbance units
  Day 1 to Day 29: number analyzed (Participants) | 32 | 32
  Day 1 to Day 29 | -2.45 (4.989) | 1.31 (10.269)
  Day 1 to Day 15 | -0.07 (4.779) | 2.55 (8.839)
  Day 29 to Day 57: number analyzed (Participants) | 31 | 31
  Day 29 to Day 57 | 3.75 (7.672) | -0.58 (10.127)

16. Other Pre Specified Outcome: Stratum Corneum Lipid Structure
Description: The difference in stratum corneum lipid structure measured by FTIR spectroscopy in conjunction with tape-stripping. FTIR spectra taken through the stratum corneum during tape-stripping on Day 29.
  Lipid chain structure was assessed by quantifying the mean frequency of the lipid peak at 2850 cm-1 (corresponding to the CH2 group of lipids). There is no range for this measurement. The higher the absorbance, the less ordered the lipid packing and weaker the structural integrity of the skin.
Time Frame: Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: absorbance units
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment
Number analyzed (Participants) | 32 | 32
absorbance units | 2849.739 (0.4140) | 2849.681 (0.4475)

17. Other Pre Specified Outcome: FLG Mutation Carriers
Description: Number of FLG loss-of-function mutation carriers
Time Frame: Saliva samples at Day 1
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 37
Participants
  wt/wt | 24
  wt/flg | 9
  wt/unknown | 4

18. Other Pre Specified Outcome: Descriptive Tabulations of TEWL by Mutation Status
Description: Descriptive tabulations of TEWL by mutation status.
Time Frame: Day 1, Day 15, Day 29 and Day 57
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: g/m²/h
Groups:
- Betamethasone Valerate (0.1%) Cream + FLG Mutation: All participants with a FLG mutation who treated with betamethasone valerate (0.1%) cream.
- Crisaborole (2%) Ointment + FLG Mutation: All participants with a FLG mutation who treated with crisaborole (2%) ointment.
- Betamethasone Valerate (0.1%) Cream Without FLG Mutation: All participants without a FLG mutation who treated with betamethasone valerate (0.1%) cream.
- Crisaborole (2%) Ointment Without FLG Mutation: All participants without a FLG mutation who treated with crisaborole (2%) ointment.
Arm/Group | Betamethasone Valerate (0.1%) Cream + FLG Mutation | Crisaborole (2%) Ointment + FLG Mutation | Betamethasone Valerate (0.1%) Cream Without FLG Mutation | Crisaborole (2%) Ointment Without FLG Mutation
Number analyzed (Participants) | 9 | 9 | 24 | 24
g/m²/h
  Day 1 | 13.7 (5.08) | 14.1 (5.94) | 13.0 (3.77) | 13.0 (4.20)
  Day 15: number analyzed (Participants) | 8 | 8 | 23 | 23
  Day 15 | 12.7 (2.86) | 15.5 (5.27) | 12.3 (2.66) | 15.0 (3.33)
  Day 29: number analyzed (Participants) | 7 | 7 | 21 | 21
  Day 29 | 11.8 (2.42) | 14.2 (5.07) | 12.5 (3.44) | 14.65 (3.48)
  Day 57: number analyzed (Participants) | 7 | 7 | 21 | 21
  Day 57 | 13.8 (3.90) | 15.2 (4.76) | 14.9 (4.26) | 15.3 (6.33)

19. Other Pre Specified Outcome: Epidermal Thickness by Mutation Status
Description: Descriptive tabulations of epidermal thickness (structural OCT derived) by mutation status.
Time Frame: Day 1, Day 15, Day 29 and Day 57.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Betamethasone Valerate (0.1%) Cream + FLG Mutation | Crisaborole (2%) Ointment + FLG Mutation | Betamethasone Valerate (0.1%) Cream Without FLG Mutation | Crisaborole (2%) Ointment Without FLG Mutation
Number analyzed (Participants) | 9 | 9 | 24 | 24
µm
  Day 1 | 101.6 (20.75) | 100.9 (17.94) | 99.4 (13.92) | 100.8 (18.39)
  Day 15: number analyzed (Participants) | 8 | 8 | 23 | 23
  Day 15 | 68.9 (11.02) | 83.5 (137.71) | 71.7 (11.25) | 86.8 (12.46)
  Day 29: number analyzed (Participants) | 7 | 7 | 21 | 21
  Day 29 | 64.4 (12.42) | 78.5 (17.96) | 67.7 (11.68) | 87.7 (12.94)
  Day 57: number analyzed (Participants) | 7 | 7 | 21 | 21
  Day 57 | 91.0 (14.47) | 100.1 (17.10) | 91.6 (9.92) | 96.0 (11.24)

ADVERSE EVENTS:
Time Frame: Incidences of adverse events were collected from the date of the first participant's enrolment (10/12/2020) until the date the last participant completed (24/09/2021). Adverse event data was collected over a period of 9 months.
Description: The definition of AE for SMART is:
  "Any untoward medical occurrence in a participant to whom a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product."
  The definition of SAE is expanded to include a point that any complications that occur during hospitalisation are to be documented as AEs. If a complication prolongs hospitalisation, this is an SAE. Elective treatment is not an AE.
Groups:
- Betamethasone Valerate (0.1%) Cream: Adverse events that can be attributed to betamethasone valerate (0.1% cream
- Crisaborole (2%) Ointment: Adverse events that can be attributed to crisaborole (2%) ointment
- Systemic Adverse Events: Adverse events that cannot be attributed to either intervention
Arm/Group | Betamethasone Valerate (0.1%) Cream | Crisaborole (2%) Ointment | Systemic Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 1/37
Other Adverse Events (participants affected / at risk) | 7/37 | 7/37 | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betamethasone Valerate (0.1%) Cream (N=37) | Crisaborole (2%) Ointment (N=37) | Systemic Adverse Events (N=37)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Abdominal and gastrointestinal infections
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betamethasone Valerate (0.1%) Cream (N=37) | Crisaborole (2%) Ointment (N=37) | Systemic Adverse Events (N=37)
Application site papules (General disorders) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 16 (16)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Thrush
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (3) | 1 (3)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Sneezing and itchy eyes
Eczema (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (5) | 2 (5)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (3) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Stomach pain
COVID-19 infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Hyperpigmentation
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site pruritis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Muscle/back pain
Application site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Trapped nerve
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Infected nail bed
Dizziness (Nervous system disorders) | 1 (2) | 1 (2) | 1 (2)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Application site rash (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT04194814/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT04194814/SAP_001.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT04194814/ICF_002.pdf